CLINICAL TRIAL: NCT01046487
Title: Imatinib Mesylate And Cyclophosphamide In Metronomic Administration: Dose Escalation Study Of Imatinib Mesylate in Patient With Rare Tumor (Phase I Study)
Brief Title: Imatinib Mesylate And Cyclophosphamide In Metronomic Administration: Dose Escalation Study Of Imatinib Mesylate
Acronym: PALANGI3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PALANGI-3 0804
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Cancer
Keywords: dermatofibrosarcoma; cylindroma; choroid melanoma; gastrointestinal stroma tumor; chordoma; ocular melanoma; conjunctival melanoma; malignant melanoma of the anus; gastric melanoma; desmoid tumor
MeSH Terms: conditions — Neoplasms; Dermatofibrosarcoma; Carcinoma, Adenoid Cystic; Uveal Melanoma; Gastrointestinal Stromal Tumors; Chordoma; Desmoid Tumors | interventions — Imatinib Mesylate; Cyclophosphamide; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Imatinib mesylate, Cyclophosphamide (Dosing level 1 ) — CYCLE 1 (42 days):
  * Day 1 to 14 Imatinib mesylate : 400 mg/day, per os
  * Day 15 to 42 Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 400 mg/day, per os
  NEXT CYCLE (28 days):
  Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 400 mg/day, per os
Drug: Imatinib mesylate, Cyclophosphamide (Dosing level 2) — CYCLE 1 (42 days):
  * Day 1 to 14 Imatinib mesylate : 600 mg/day,(300 mg in the morning and 300 mg in the evening) per os
  * Day 15 to 42 Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 600 mg/day,(300 mg in the morning and 300 mg in the evening) per os
  NEXT CYCLE (28 days):
  Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 600 mg/day,(300 mg in the morning and 300 mg in the evening)per os
Drug: Imatinib mesylate, Cyclophosphamide (Dosing level 3) — CYCLE 1 (42 days):
  * Day 1 to 14 Imatinib mesylate : 800 mg/day,(400 mg in the morning and 400 mg in the evening) per os
  * Day 15 to 42 Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 800 mg/day,(400 mg in the morning and 400 mg in the evening) per os
  NEXT CYCLE (28 days):
  Cyclophosphamide : 50 mg x 2/day, per os Imatinib mesylate : 800 mg/day,(400 mg in the morning and 400 mg in the evening)per os
Procedure: Blood sampling — ONLY FOR CYCLE 1, at day 15 and day 28 :
  11 sampling for dosing level 1 (pre-dose, imatinib mesylate + 30 min, +1, +2, +3, +4, +6, +10, +12 , +24 hours, cyclophosphamide + 12 hours) 10 sampling for the next dosing level (pre-dose, imatinib mesylate + 30 min, +1, +2, +3, +4, +6, +10, +12,cyclophosphamide + 12 hours)

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of imatinib mesylate, given in association with a fixed dose of cyclophosphamide (50 mg bid).

ELIGIBILITY:
Inclusion Criteria:

* Rare tumor
* metastatic disease or locally advanced disease, inoperable, with no standard treatment
* At least 28 days since the prior treatment
* Measurable disease with at least one measurable lesion

Exclusion Criteria:

* Medullary insufficiency
* Cystitis, haemorrhagic cystitis
* Hepatic porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
For safety: NCI-CTCAE scale version 3.0 | 42 days

SECONDARY OUTCOMES:
For anti tumoral efficiency : RECIST criteria | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (3):
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon